CLINICAL TRIAL: NCT02016859
Title: Observational Prospective Study of the Predicted Value of Immature Thrombocytes Counts in Three Different Groups of Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Yishai Ofran (Other)
Responsible Party: Sponsor-Investigator, Dr. Yishai Ofran, Doctor, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Other Study IDs: IPF-2013-Rambam
Record Dates: First submitted 2013-11-10; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Critically Ill Patients; Neutropenic Fever Patients; Patients With Hip Fractures
Keywords: IPF Immature platelet fraction; ICU neutropenic fever; hip fracture; critically ill
MeSH Terms: conditions — Hip Fractures; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Critically ill patients admitted to ICU: those patients who are admitted to ICU with multiorgan failure/injury
  Interventions: Other: Immature Platelet Fraction
- Neutropinc Fever patients: admitted to ER, haemato-oncology or oncology
  Interventions: Other: Immature Platelet Fraction
- Patients of Hip's Fracture: admitted to orthopedic departement
  Interventions: Other: Immature Platelet Fraction

INTERVENTIONS:
Other: Immature Platelet Fraction

SUMMARY:
Immature Platelet Fraction (IPF) is a new value in CBC blood tests Recent Studies showed that this value may be another prognostic factor in critically ill patients such as those admitted to ICU, or those with neutropenic Fever.

The purpose of the study is to check if the IPF may be used as a prognostic Factor in these patients

DETAILED DESCRIPTION:
In this study we have 3 groups of patients

* Patients admitted to ICU
* Patients admitted with neutropenic fever
* Patients admitted with hip fractures it is a prospective study, not interventional, we'll take blood samples of these patients including CBC count eith IPF and other inflammation markers such as CRP and we'll compare CRP to IPF in addition to clinical follow-up of the patient till discharge.

At the end of this study we'll compare the efficacy of IPF as a prognostic Factor in these patients

ELIGIBILITY:
Inclusion Criteria:

- Admission to hospital blood sample is taken between 24:00 pm till 15:00 pm

Exclusion Criteria:

* blood sample is taken after 15:00 pm in the first day of admission during the week
* blood sample is taken on weekend: thursday 15:00 pm till saturday 24:00 pm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: admmitted patients to multiple departements
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-05 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Time to recovery from sepsis or time to death | 6 months
  the primary outcome is the result of the patient's admission on which data analysis will be based

SECONDARY OUTCOMES:
Predicting value of IPF for prognosis | baeline 6 months
  after the analysis of the data we'll may ba able to assess the predicting value of the IPF in predicting severity of infection and prediciting prognosis of infection in the three groups described

OTHER OUTCOMES:
clinical use of IPF as a prognostic factor | up to 12 months
  this outcome is not uet based we need much more studies in order to be able to use IPF in daily clinical work

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health care campus, Haifa, Israel

REFERENCES:
- [Result] Di Mario A, Garzia M, Leone F, Arcangeli A, Pagano L, Zini G. Immature platelet fraction (IPF) in hospitalized patients with neutrophilia and suspected bacterial infection. J Infect. 2009 Sep;59(3):201-6. doi: 10.1016/j.jinf.2009.07.007. Epub 2009 Jul 18. PMID 19647322
- [Result] De Blasi RA, Cardelli P, Costante A, Sandri M, Mercieri M, Arcioni R. Immature platelet fraction in predicting sepsis in critically ill patients. Intensive Care Med. 2013 Apr;39(4):636-43. doi: 10.1007/s00134-012-2725-7. Epub 2012 Oct 24. PMID 23093245